CLINICAL TRIAL: NCT06486961
Title: Randomized Controlled Study of the Effectiveness of a Self-rehabilitation Program for Walking Using Adapted Musical Auditory Rhythmic Stimulation, Delivered by BeatMove, in People Suffering From Obesity
Brief Title: Effect of Walking With Music in Obese People (BeatMove)
Acronym: BeatMove
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Beau Soleil (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-A01544-39
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Sedentary Behavior
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BeatMove Experimental Group (Experimental): The participant walks for 15 to 30 minutes a day, 5 day a week for 3 months. During the walking session, BeatMove application delivers synchronized music adapted to the patient walking.
  The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Interventions: Device: BeatMove Application
- Control Group with Music at Random Tempo (Active Comparator): The participant walks for 15 to 30 minutes a day, 5 day a week for 3 months. During the walking session, BeatMove Application delivers random music at random tempo.
  The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Interventions: Device: BeatMove Application without synchronized music
- Control Group without Music (Active Comparator): The participant walks for 15 to 30 minutes a day, 5 day a week for 3 months. During the walking session, BeatMove Application does not deliver music. The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Interventions: Device: BeatMove Application without music

INTERVENTIONS:
Device: BeatMove Application — The participant walks for 15 to 30 minutes a day, 5 day a week for 3 months. During the walking session, BeatMove application delivers synchronized music adapted to the patient walking.
  The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Arms: BeatMove Experimental Group
Device: BeatMove Application without synchronized music — The participant walks for 15 to 30 minutes a day, 5 day a week for 3 months. During the walking session, BeatMove Application delivers random music at random tempo.
  The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Arms: Control Group with Music at Random Tempo
Device: BeatMove Application without music — The participant walks for 15 to 30 minutes a day, 5 day a week for 3 months. During the walking session, BeatMove Application does not deliver music. The application allows participants to know the progress of their session through graphical representation and voice messages, informs them at the end of the session of their performance and congratulate them for their efforts.
  Arms: Control Group without Music

SUMMARY:
For several decades, scientists have reported encouraging effects of physical activity on functional capacities and quality of life among patients with obesity. However, regular daily physical activity remains limited in these individuals. People with obesity generally show lower adherence to physical activity, with 40% not meeting the recommendations of 2.5 to 3 hours of moderate physical activity per week set by the French National Authority for Health to be considered physically active. Since physical activity is the primary energy expenditure that can be targeted, the priority is to make it appealing through exercise programs tailored to individual needs, abilities, and preferences. To achieve this, using music to facilitate walking appears relevant. Studies show that individuals adhere to physical activity and incorporate it into their routines only if they find it enjoyable. Walking to music is more motivating and enjoyable. Moreover, the rhythm of music enhances the functioning of biological systems involved in walking. Tailored physical activity is a major preventive lever to implement for individuals with obesity. It is essential during the initial weight loss phase and during weight maintenance.

The overall objective of this study is to propose a digital tool capable of modifying the behavior of individuals with obesity to reduce sedentary behavior in their daily lives. Synchronized walking to the rhythm of music should help train obese patients towards a virtuous cycle leading to slowed weight gain, reduced associated health problems, and improvements in mental health and quality of life.

DETAILED DESCRIPTION:
This program involves outdoor walking sessions, conducted 5 times a week for 15 to 30 minutes each, over a consecutive 3-month period using the BeatMove device. The device can be adjusted to deliver music or not, and the music can either be synchronized to the participant's walking pace or randomly timed.

During the week preceding self-rehabilitation, participants will wear a thigh-mounted accelerometer to establish a baseline representative of their daily habits. Before each walking session, participants will assess their motivation using a visual analog scale within the application. After each session, they will evaluate their perceived exertion using the Borg Scale.

In the BeatMove group, the music delivered will be tailored to match the walking pace of the participants. Throughout the session, the music rhythm will subtly increase by 20% to accelerate the participant's walking pace, thereby guiding them towards their optimal cadence based on their assessed level and motivation at the start of the session.

In the group with randomly timed music, the music delivery does not consider the participant's state and plays random music.

Finally, in the group without music, the walking self-rehabilitation program will be guided solely by the audio instructions provided by the application.

In all three groups, participants will be equipped:

Throughout the day with a thigh-mounted "fibion sens" accelerometer. During the walking self-rehabilitation session with ankle step sensors to record walking parameters while delivering music tailored to their walking pace.

ELIGIBILITY:
Inclusion Criteria:

* Be able to walk continuously for 15 minutes without the use of any assistive devices (e.g., cane, walker) or human assistance.
* Have a Body Mass Index (BMI) greater than 25 and less than 45.
* Understand the nature, purpose, and methodology of the study.
* Agree to cooperate during evaluations.
* Have signed the informed consent form.
* Be affiliated with a social security scheme or equivalent.

Exclusion Criteria:

* Marcher plus de 30 minutes, 5 fois par semaine
* Présenter une insuffisance cardiaque ou respiratoire sévère contre indiquant une rééducation à la marche.
* Majeurs faisant l'objet d'une protection légale ou hors d'état d'exprimer leur consentement (Article 1121-8 du CSP)
* Personnes vulnérables (Article L 1121-6 du CSP)
* Privation de liberté par décision judiciaire ou administrative
* Forte probabilité de non-compliance au protocole ou d'abandon en cours d'étude
* Femmes enceintes/allaitantes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Differences in average daily step count | Up to 3 months
  The primary outcome measure is the variation in average daily step count across the three groups during the week (7 consecutive days) prior to the start of home-based self-rehabilitation and the final week of self-rehabilitation. These steps will be measured using "fibion sens" accelerometers under ecological conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Attalin, Dr, Principal Investigator — Clinique Beau Soleil
Locations (1):
- Clinique Beau Soleil, Montpellier, Hérault, France